CLINICAL TRIAL: NCT00651651
Title: A 12 Week Randomized, Double-blind, Double-Dummy, Placebo-controlled Trial of Symbicort TM (160/4.5mcg) Versus Its Mono-Products (Budesonide and Formoterol) in Children (at Least 6years of Age) and Adults With Asthma-SPRUCE 80/4.5
Brief Title: Efficacy of Symbicort Versus Its Monocomponents - SPRUCE 80/4.5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SD-039-0716; D5896C00716
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Symbicort; budesonide/formoterol; budesonide; formoterol
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Symbicort
  Interventions: Drug: budesonide/formoterol
- 2 (Active Comparator): budesonide
  Interventions: Drug: budesonide
- 3 (Active Comparator): formoterol
  Interventions: Drug: formoterol

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: budesonide
  Arms: 2
Drug: formoterol
  Arms: 3

SUMMARY:
The purpose of this study is to compare Symbicort with its monocomponents budesonide and formoterol in the treatment of asthma in children and adults

ELIGIBILITY:
Inclusion Criteria:

* At least 6 years of age
* Diagnosis of asthma
* Baseline lung function test results as determined by protocol and required and received treatment with inhaled corticosteroids and/or lung treatments specified in protocol within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Severe asthma
* Has required treatment with any non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers
* Had cancer within previous 5 years or currently has any other significant disease or disorder as judged by the investigator

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2002-08; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
12 hour serial FEV1 measurements and withdrawals due to asthma exacerbation | FEV1: before start of tretment and at 2 and 12 weeks after start of treatment. Withdrawals: throughout the treatment period

SECONDARY OUTCOMES:
Lung function, asthma symptoms, use of rescue medication, adverse events and other safety assessments | Throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca

REFERENCES:
- [Derived] Murphy KR, Uryniak T, Martin UJ, Zangrilli J. The effect of budesonide/formoterol pressurized metered-dose inhaler on predefined criteria for worsening asthma in four different patient populations with asthma. Drugs R D. 2012 Mar 1;12(1):9-14. doi: 10.2165/11630600-000000000-00000. PMID 22329608